CLINICAL TRIAL: NCT05213572
Title: Observational Study to Deeply Phenotype Major Organs in Sickle Cell Disease After Curative Therapies
Status: Recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000479; 000479-H
Record Dates: First submitted 2022-01-27; First posted 2022-01-28 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11-06

CONDITIONS: Mortality in Sickle Cell; Sickle Cell Cardiopulmonary Complications; Sickle Cell Organ Damage; Sickle Cell Life Expectancy and Risk Factors for Early Death; Sickle Cell Lung Disease and Sudden Death
Keywords: Hydroxyurea; Hydroxyurea-Increased Fetal Hemoglobin; sickle cell anemi; Patterns of mortality in sickle cell disease; Mortality rates and age at death from sickle cell; Natural History
MeSH Terms: conditions — Death, Sudden

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- subjects w sickle cell disease: to evaluate heart, lung, liver, kidney, brain, and neurocognitive function post-hematopoietic stem cell transplant (HSCT) in subjects with sickle cell disease (SCD) who undergo curative therapies

SUMMARY:
Background:

People with sickle cell disease (SCD) have problems with their heart, brain, kidneys, liver, and lungs as they age. These problems may improve after transplant. Researchers want to learn how and why this happens.

Objective:

To study the benefits of treatments that are intended to cure SCD.

Eligibility:

People aged 18 and older with SCD who are either receiving curative therapy in the next 3 months or don t have any plans to receive a curative therapy in the next 2 years.

Design:

At their first visit, participants will be screened with their medical history and a physical exam.

Participants will then have a baseline visit. This will take about a week to complete and will include:

Blood and heart tests

MRI of the brain, heart, and lungs. Participants will lie on a bed that will move into the MRI scanner. Special padding may be placed around their head to keep it still.

Interactive games. Participants will complete computer games that test memory, attention, problem solving, language, spatial orientation, processing speed, and emotion.

Questionnaire rating quality of life

Iothalamate test. An IV catheter will be placed into a vein. A contrast agent will be injected through the IV. Blood will then be collected at different time points.

Lung function tests and a 6-minute walk test

Vibration controlled transient elastography. A probe placed on the abdomen will measure liver scarring.

DOS test. A light attached to the finger or toe will measure blood oxygen.

Participants will have an end-of-study visit about 2 years after their baseline visit. This will include repeats of the baseline visit tests.

DETAILED DESCRIPTION:
Study Description:

This study seeks to evaluate heart, lung, liver, kidney, brain, and neurocognitive function post-hematopoietic stem cell transplant (HSCT) in patients with sickle cell disease (SCD) who undergo curative therapies. Based on our preliminary data, the primary hypothesis is that diastolic function will improve after successful curative therapy as compared to baseline. Secondary analyses will include assessment of cardiopulmonary and kidney function. This study includes assessment of organs before and 2 years after curative therapies with deep phenotyping of the heart, lung, liver, brain, cognitive, and kidney function. Patients who undergo curative therapies will be compared to adults with SCD who receive non-curative therapies at baseline and 2 years later. This protocol will allow us to comprehensively explore sequelae of curative therapies on organ function in patients with SCD.

Objectives:

Primary Objective:

-Evaluate left ventricular end diastolic volume/body surface area (LVEDV/BSA) in patients with SCD who undergo curative therapies as compared to patients who receive non-curative therapies at 2 years after initial testing.

Secondary Objectives:

* Evaluate other markers of cardiopulmonary function in patients with SCD who undergo curative therapies as compared to those who receive non-curative therapies.
* Evaluate change in kidney function over time in patients with SCD who undergo curative therapies as compared to those who receive non-curative therapies.

Tertiary Objectives:

* Perform deep phenotyping of heart, lung, liver, kidney, brain and neurocognitive function along with reported genetic variants in adults with SCD who undergo curative therapies as compared to adults with SCD who receive non-curative therapies.
* Assess markers of inflammation in patients with SCD who undergo curative therapies as compared to those who receive non-curative therapies.
* Evaluate markers of graft rejection and tolerance induction in patients with SCD who undergo curative therapies.
* Evaluate lipid profiles in patients with SCD who undergo curative therapies as compared to those who receive non-curative therapies.
* Evaluate regional oxygenation (rS02) with Near Infrared Spectroscopy (NIRS) in patients with SCD who undergo curative therapies as compared to those who receive non-curative therapies.
* Evaluate novel biomarkers of organ damage in patients who receive curative therapies as compared to those who receive non-curative therapies.

Endpoints:

Primary Endpoint:

-Change in LVEDV/BSA

Secondary Endpoints:

* Change in left ventricular end diastolic diameter (LVEDD), ejection fraction, left ventricular mass index, left atrial volume index, global longitudinal strain
* Change in N-terminal pro b-type natriuretic peptide (NTproBNP).
* Change in creatinine, cystatin-C, urine protein to creatinine ratio, urine albumin to creatinine ratio, and estimated glomerular filtration rate (eGFR) using the CKD-EPI equation

Tertiary Endpoints:

* Change in myocardial fibrosis, extracellular volume fraction, processing speed, measured GFR, incidence of stroke/silent infarcts, cerebral blood flow, oxygen extraction fraction, and liver stiffness, and correlation of APOL1 risk alleles with renal function and degree of proteinuria
* Change in c-reactive protein (CRP), erythrocyte sedimentation rate (ESR), inflammatory cytokines (including interferon gamma (IFN-y) and tumor necrosis factor alpha (TNF-a), chemokines, GlycA, D-dimer, and haptoglobin
* Change in regulatory cells (including regulatory T cells and myeloid-derived suppressor cells) and proteins (including galectin, platelet factor 4, and thrombospondin-1) and suppressive cytokines (interleukin-10 (IL-10), transforming growth factor beta, and IL-7)
* Change in very low-density lipoprotein (VLDL), low-density lipoprotein (LDL) and high-density lipoprotein (HDL) particle size and number, triglycerides, and apolipoprotein A-I and B
* Change in rS02 within the peripheral limb with NIRS
* Correlation of novel genetic biomarkers associated with organ damage in patients with SCD who receive curative therapy or noncurative therapy.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study
2. Male or female, aged >=18 years
3. Current or previous diagnosis of any type of SCD (including HbSS, HbSC, HbSbeta0-thal, HbSbeta+-thal)
4. Ability to travel to the NIH Clinical Center
5. Ability of subject to understand and the willingness to sign a written informed consent document.
6. Ability to undergo required studies except as specified in the Exclusion Criteria.
7. Curative Therapies Group

   --Plan to receive conditioning for curative therapy at the NIH Clinical Center, Vanderbilt University Medical Center, or Johns Hopkins Hospital
8. Non-Curative Therapy Group

   -- No plan to undergo curative therapy within 2 years
9. At least one of the following eligibility criteria:

   * History of stroke or abnormal transcranial doppler examination (>= 200 m/s)
   * History of SCD-related renal insufficiency defined as a creatinine level >=1.3 mg/dL and kidney biopsy consistent with sickle cell nephropathy OR nephrotic syndrome OR creatinine clearance < 50mL/min
   * Tricuspid regurgitant velocity >= 2.5 m/s
   * Recurrent tricorporal priapism defined as at least 2 episodes of an erection lasting > 4 hours involving the corpora cavernosa and corpus spongiosa
   * SCD-associated liver disease defined as EITHER ferritin > 1000 mcg/L OR direct bilirubin > 0.4 mg/dL
   * > 1 hospitalization per year for vaso-occlusive crises while on a therapeutic dose of hydroxyurea
   * Any acute chest syndrome while on a therapeutic dose of hydroxyurea
   * Osteonecrosis of 2 or more joints
   * Red cell alloimmunization

EXCLUSION CRITERIA:

All individuals meeting any of the exclusion criteria at baseline will be excluded from study participation.

1. Prior transplantation (including but not limited to HSCT and kidney transplant)
2. Pregnant or breastfeeding
3. Patients with allergy to iodine or iodinated contrast solutions will not undergo Iothalamate or Iohexal GFR clearance testing but can undergo the other deep phenotype testing
4. Implanted metal object that is not compatible with MRI (e.g.: cerebral aneurysm clip, cochlear implant, or pacemaker)
5. Patients with a pacemaker or automated implantable cardioverter defibrillator will not undergo VCTE but can enroll and undergo the other deep phenotype testing as long as the device is compatible with MRI and MRI testing can be performed
6. Patients requiring peritoneal or hemodialysis
7. Uncontrolled infection or acute illness
8. Criteria specific to the non-curative therapy group:

   1. Hydroxyurea initiation or dose adjustment <2 months prior
   2. Initiation of chronic transfusion therapy <2 months prior
   3. Antihypertensive medication initiation or dose adjustment <1 month prior

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged >or= 18 years who will undergo curative therapies at the NIH Clinical Center and who have a diagnosis of any type of SCD (including HbSS, HbSC, HbSbeta0-thal, HbSbeta+-thal).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-03-24 (Actual); Primary Completion 2035-06-01 (Estimated); Study Completion 2035-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in LVEDV/BSA in patients with SCD who undergo curative therapies as compared to patients who receive non-curative treatment | 2 years after initial testing
  Evaluate whether diastolic function improves significantly more in patients who receive curative therapies as compared to those who receive non-curative treatment.

SECONDARY OUTCOMES:
Change in creatinine, cystatin-C, urine protein to creatinine ratio, urine albumin to creatinine ratio, and estimated glomerular filtration rate (eGFR) using the CKD-EPI equation | 2 years
  Evaluate change in kidney function over time in patients with SCD who undergo curative therapies as compared to those who receive non-curative treatment.
Change in N-terminal pro b-type natriuretic peptide (NTproBNP). | 2 years
  Evaluate whether cardiopulmonary function improves more in patients who receive curative therapies as compared to non-curative therapy.
Change in left ventricular end diastolic diameter (LVEDD), ejection fraction, left ventricular mass index, left atrial volume index, global longitudinal strain | 2 years
  Evaluate whether cardiopulmonary function improves more in patients who receive curative therapies as compared to non-curative therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney F Joseph, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000479-H.html